CLINICAL TRIAL: NCT00026195
Title: Clinical Pharmacology In The Elderly: Prospective Evaluation Of The Pharmacokinetics, Pharmacogenetics And Pharmacodynamics Of CPT-11 And Aging
Brief Title: Irinotecan in Treating Aging Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-60001; U10CA031946 (NIH); CLB-60001; CDR0000068995 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- irinotecan (Experimental): Patients receive irinotecan IV over 90 minutes once weekly for 4 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Patients are followed for survival.
  Interventions: Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Aging may affect the way these drugs work.

PURPOSE: Phase I trial to determine the relationship between aging and the effectiveness of irinotecan in treating patients who have solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether there is a relationship between the pharmacokinetic characteristics of irinotecan and aging in patients with non-hematologic malignancies.
* Determine whether there is a relationship between the toxic effects of this drug and aging in these patients.
* Determine whether the relationship between genotype (UGT1A1, CYP3A, and other relevant genes) and phenotype (pharmacokinetics, toxicity) is affected by aging in these patients treated with this drug.
* Analyze data collected on the co-morbid conditions and concurrent medications in these patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to age (18 to 55 vs 70 and over).

Patients receive irinotecan IV over 90 minutes once weekly for 4 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 140 patients (70 per stratum) will be accrued for this study within 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-hematologic malignancy
* Brain metastases or primary brain tumors are eligible provided patient is not receiving steroids or antiepileptic medications

PATIENT CHARACTERISTICS:

Age:

* 18 to 55 or 70 and over

Performance status:

* CTC 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* SGOT no greater than ULN

Renal:

* Creatinine no greater than ULN

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosourea)
* No more than 1 prior chemotherapy regimen for metastatic disease (no limit if administered in the adjuvant setting)
* No prior camptothecin

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy, including for palliation

Surgery:

* At least 4 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2001-09; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
overall survival | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M. Lichtman, MD, Study Chair — Don Monti Comprehensive Cancer Center at North Shore University Hospital
Locations (47):
- United States (47):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - MBCCOP - Massey Cancer Center, Richmond, Virginia